CLINICAL TRIAL: NCT00415818
Title: A Phase IIb Multicentric Controlled Study Evaluating the Therapeutic Vaccine TG4010(MVA-MUC1-IL2) as an Adjunct to Standard Chemotherapy in Advanced Non Small Cell Lung Cancer
Brief Title: Immunotherapy With TG4010 in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Transgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG4010.09
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung Cancer; NSCLC; Cancer Vaccine; Stage IV Non-Small Cell Lung Cancer; Stage IIIb Non-Small Cell Lung Cancer with effusion
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

ARMS (2):
- Arm 1 (Experimental): MVA-MUC1-IL2 in combination with 1st line Chemotherapy
  Interventions: Biological: MVA-MUC1-IL2; Drug: 1st line Chemotherapy
- Arm 2 (Active Comparator): 1st line Chemotherapy without a MVA-MUC1-IL2 combination
  Interventions: Drug: 1st line Chemotherapy

INTERVENTIONS:
Biological: MVA-MUC1-IL2 — MVA-MUC1-IL2:
  Dose of 10exp8 plaque forming units (pfu).
  Chemotherapy:
  Arm 1 and Arm 2 Intravenous CT: cisplatin (75mg/m² at Day 1) and gemcitabine (1250mg/m² at Days 1 and 8) every 3 weeks, for up to six cycles or until progressive disease, whichever occurred first.
  Arms: Arm 1
Drug: 1st line Chemotherapy

SUMMARY:
The primary Objective is to assess the efficacy of TG4010 combined to chemotherapy in comparison with chemotherapy alone in patients with advanced non small cell lung cancer.

DETAILED DESCRIPTION:
In the experimental arm patients receive subcutaneous injections of TG4010 at the dose of 108 pfu in combination with chemotherapy treatment whereas patients in the control arm receive chemotherapy alone. The chemotherapy associates cisplatin and gemcitabine and is given for up to 6 cycles or progressive disease, whichever occurs first.

TG4010 is administered once per week for 6 weeks, then once every 3 weeks in combination with chemotherapy and thereafter as monotherapy until documentation of progressive disease.

Tumor response will be evaluated every 6 weeks by a CT-scan and results will be available before starting an additional treatment period of 6 weeks. The tumor response taken into account will be for each patient the best overall response obtained during the study.

The endpoint of the study is based on Progression Free Survival (PFS) at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell carcinoma of the lung (adenocarcinoma, squamous cell carcinoma, or large cell carcinoma);
* Histological documentation of MUC1 antigen expression on the primary tumor or on metastasis, as defined by a positive staining by immuno-histo-chemistry in at least 25% of the tumor cells in the conditions described in the technical documentation of the monoclonal antibody;
* Patients will have stage IIIb "wet" (with pleural or pericardial effusion) or IV disease, with no prior systemic therapy for advanced disease except for adjuvant treatment. Prior surgery or radiation therapy aimed at local palliation or attempted local disease control is permitted;
* At least one measurable lesion by Computed Tomography (CT-scanner) according to WHO criteria (lesion accurately measured in two dimensions with longest diameter equal or greater to 10 mm with spiral CT scan);
* Adequate hematological, hepatic, and renal function:

  * Hemoglobin >= 10.0 g/dL; WBC >= 3.0x10e9/L including neutrophils >= 1.5x10e9/L and total lymphocytes count >= 0.5x10e9/L; platelets count >= 100x10e9/L;
  * Bilirubin =< 2x the upper limit of normal and serum transaminases =< 3x the upper limit of normal;
  * Glomerular Filtration Rate higher than 60 ml/mn according to Cockcroft formula;
* Performance status 0 or 1 on the ECOG scale (Appendix 2);
* Minimum estimated life expectancy of 4 months;
* Written informed consent from patient.

Exclusion Criteria:

* Concomitant brain metastases. If previous brain metastases were treated, the absence of evolution is to be demonstrated by the MRI or scanner performed at baseline;
* Prior history of other malignancy except basal cell carcinoma and intra-epithelial cervical cancer or other cancer with complete response since at least 5 years;
* History of any form of systemic therapy for advanced non-small cell cancer of the lung except for (neo)adjuvant treatment;
* Previous (within 4 weeks prior to day 1) or concomitant long term treatment with systemic steroids, immunosuppressive / immunomodulating drugs (e.g. Cyclosporine, corticoïds);
* Positive serology for HIV or HCV; positive antigens for hepatitis B;
* Serious concomitant medical disorder;
* Major surgery within 4 weeks prior to day 1;
* Patient with an organ allograft;
* Allergy to eggs;
* Participation in another experimental protocol during the study period, or within 4 weeks prior to day 1;
* Pregnancy at the entry or women who are breast feeding;
* Patient without adequate protection against pregnancy during the conduct of the study and for 3 months after the last injection of TG4010 and/or chemotherapy;
* History of substance abuse;
* Patient unable or unwilling to comply with the protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2005-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Progression free survival at 6 months | 6 months

SECONDARY OUTCOMES:
Response Rate according to WHO criteria | 6 months
Time to progression | 6 months
Overall survival
Quality of life | every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth QUOIX, M.D., Principal Investigator — Hôpital Lyautey, Service de Pneumologie
Locations (23):
- France (11):
  - Centre Hospitalier Belfort-Montbeliard, Belfort
  - CHU, Service de Pneumologie, Besançon
  - Centre Hospitalier Général, Service de Pneumologie, Briey
  - Centre François Baclesse, Caen
  - Hôpital Pasteur - Service de médecine F- Pavillon 43, Colmar
  - Centre Oscar Lambret, Lille
  - Institut Paoli-Calmettes, Service d'oncologie médicale, Marseille
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHRU Hôpital de Pontchaillou, Rennes
  - Hôpital Lyautey - Service de Pneumologie, Strasbourg
  - Centre Hospitalier de la Haute Saône, Service de Pneumologie - Allergologie, Vesoul
- Germany (5):
  - Lungenklinik Krankenhaus Merheim, Cologne
  - Asklepios Fachkliniken, Zentrum für Pneumonologie, Gauting
  - Thoraxklinik Heidelberg, Heidelberg
  - Klinikum Mannheim der Ruprecht-Karls, Mannheim
  - Klinikum Offenburg, Medizinische Klinik II, Offenburg
- Fejér Megyei Szent György Kórház, Székesfehérvár, Hungary
- Poland (6):
  - Oddział II Chorób Płuc i Gruźlicy, Bialystok
  - Kujawsko-Pomorskie Centrum Pulmonologii, Bydgoszcz
  - Oddział Chemioterapii, Krakow
  - Oddział III Chorób Płuc i Gruźlicy, Otwock
  - Oddział Onkologii Klinicznej, Poznan
  - Dolnośląskie Centrum, Wroclaw

REFERENCES:
- [Result] Quoix E, Ramlau R, Westeel V, Papai Z, Madroszyk A, Riviere A, Koralewski P, Breton JL, Stoelben E, Braun D, Debieuvre D, Lena H, Buyse M, Chenard MP, Acres B, Lacoste G, Bastien B, Tavernaro A, Bizouarne N, Bonnefoy JY, Limacher JM. Therapeutic vaccination with TG4010 and first-line chemotherapy in advanced non-small-cell lung cancer: a controlled phase 2B trial. Lancet Oncol. 2011 Nov;12(12):1125-33. doi: 10.1016/S1470-2045(11)70259-5. Epub 2011 Oct 21. PMID 22019520
- See also: Related Info — http://www.nlm.nih.gov/medlineplus/lungcancer.html